CLINICAL TRIAL: NCT00000842
Title: A Phase II, Double-Blind Trial of Recombinant Human Nerve Growth Factor for Treatment of HIV-Associated Sensory Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 291; 11267 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Peripheral Nervous System Disease
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Peripheral Nervous System Diseases; Nerve Growth Factors; Growth Substances
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nerve Growth Factor

INTERVENTIONS:
Drug: Nerve Growth Factor, Recombinant Human

SUMMARY:
To assess the efficacy, safety, and tolerability of recombinant human nerve growth factor ( rhNGF ) in the treatment of HIV-associated sensory neuropathy. AS PER AMENDMENT 5/6/97: To compare the change in viral load between the double-blind phase baseline and week 4 in placebo and active rhNGF recipients. To ensure that rhNGF does not induce an increase in viral load compared with viral load changes seen with placebo.

Up to now, treatments for HIV-associated sensory neuropathy have been symptomatic, relying on pain-modifying agents or membrane-stabilizing drugs. Because nerve growth factor is important in the development and maintenance of sympathetic and sensory neurons and their outgrowths, it is proposed that recombinant human nerve growth factor may provide a specific restorative treatment for HIV-associated painful sensory neuropathy.

DETAILED DESCRIPTION:
Up to now, treatments for HIV-associated sensory neuropathy have been symptomatic, relying on pain-modifying agents or membrane-stabilizing drugs. Because nerve growth factor is important in the development and maintenance of sympathetic and sensory neurons and their outgrowths, it is proposed that recombinant human nerve growth factor may provide a specific restorative treatment for HIV-associated painful sensory neuropathy.

Patients are randomized to receive either rhNGF at one of two doses or placebo, administered subcutaneously twice weekly for 18 weeks. Patients are stratified into three groups within their regimens by use of didanosine, zalcitabine, or stavudine as follows: current use vs. discontinued between 8 and 26 weeks before randomization vs. never used or discontinued use at least 26 weeks before randomization. Patients will assess their pain daily using the Gracely Pain Scale. AS PER AMENDMENT 5/6/97: After completion of the double-blind phase (18 weeks on treatment followed by 4 weeks off treatment), patients may receive open-label, active drug treatment according to their previously assigned regimen for an additional 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Maintenance treatment of CMV retinitis, MAI bacteremia, or cryptococcal meningitis is permitted.
* Local therapy for Kaposi's sarcoma.

Patients must have:

* Evidence of HIV antibodies documented by a licensed ELISA and a second, FDA-approved, confirmatory test.
* Diagnosis of HIV-associated, predominantly sensory neuropathy by a neurologist.
* Willingness and ability to complete the pain and medication log and competence to assess pain level throughout the study.

Prior Medication:

Allowed:

* History of stable-dose (defined as no more than 50% increase or decrease in dose) antiretroviral therapy for eight weeks before randomization, including the following:
* didanosine, zalcitabine, stavudine, lamivudine, protease inhibitors, and antiretrovirals available through expanded access trials.
* Chemotherapeutic drugs other than neurotoxic systemic chemotherapeutic agents within 30 days prior to randomization.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Presence of acute, active, opportunistic infection, except oral thrush; oral, genital or rectal herpes; and MAI bacteremia within two weeks before randomization.
* Evidence of another contributing cause for peripheral neuropathy, including:
* diabetes mellitus, hereditary neuropathy, current vitamin B12 deficiency and no supplementation or supplementation <= 3 months, or treatment with any drug that might contribute to sensory neuropathy.
* Major active psychiatric disorder (depression is allowed provided patient has received a stable antidepressant regimen for at least four weeks before randomization).
* Current active malignancy. NOTE: Malignancies in remission that do not require further treatment or Kaposi's sarcoma requiring only local treatment are allowed.
* Any conditions, including dementia and myelopathy, that would interfere with patient evaluation, accurate completion of the symptom scale, or compliance with subcutaneous injection.

Concurrent Medication:

Excluded:

* Chemotherapeutic agents.
* Systemic corticosteroids or immunomodulators.
* Initiation of new antiretroviral to a stable regimen.

Prior Medication:

Excluded:

* Neurotoxic systemic chemotherapy within the past 90 days.
* Systemic corticosteroids or immunomodulators within the past 30 days.
* Initiation of non-opioid prescription medication for pain during the 2 weeks preceding randomization (including tricyclic antidepressants, mexiletine, phenytoin, and carbamazepine).
* Treatment for acute opportunistic infections within the past 14 days (maintenance therapy for CMV retinitis, MAI bacteremia, or cryptococcal meningitis is permitted).

Active drug or alcohol abuse that would affect study compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Study Completion 1999-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McArthur J, Study Chair; Simpson D, Study Chair; Schifitto G, Study Chair
Locations (14):
- United States (14):
  - UCLA CARE Center CRS, Los Angeles, California
  - San Mateo County AIDS Program, San Mateo, California
  - Stanford CRS, Stanford, California
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Nerve growth factor study opens. GMHC Treat Issues. 1996 Nov;10(11):9. PMID 11364013
- [Background] Gilden D. Hyperthermia study finds little effect. GMHC Treat Issues. 1995 Nov;9(11):5-7. PMID 11362992
- [Background] James JS. Nerve growth factor: major trial canceled, revived after protest. AIDS Treat News. 1995 Apr 21;(no 221):5. PMID 11362404
- [Background] Simpson DM, Haidich AB, Schifitto G, Yiannoutsos CT, Geraci AP, McArthur JC, Katzenstein DA; ACTG 291 study team. Severity of HIV-associated neuropathy is associated with plasma HIV-1 RNA levels. AIDS. 2002 Feb 15;16(3):407-12. doi: 10.1097/00002030-200202150-00012. PMID 11834952
- [Background] Lein B. Potential therapy for painful neuropathy. PI Perspect. 1995 May;(no 16):11. PMID 11362419
- [Background] McArthur JC, Yiannoutsos C, Simpson DM, Adornato BT, Singer EJ, Hollander H, Marra C, Rubin M, Cohen BA, Tucker T, Navia BA, Schifitto G, Katzenstein D, Rask C, Zaborski L, Smith ME, Shriver S, Millar L, Clifford DB, Karalnik IJ. A phase II trial of nerve growth factor for sensory neuropathy associated with HIV infection. AIDS Clinical Trials Group Team 291. Neurology. 2000 Mar 14;54(5):1080-8. doi: 10.1212/wnl.54.5.1080. PMID 10720278